CLINICAL TRIAL: NCT03259932
Title: Personalised Physical Training Associated With Usual Management Versus Usual Management Alone on Fatigue and Recovery After Minor Stroke: Randomised Controlled Trial
Brief Title: Comparison of Fatigue and Recovery After Stroke Depending on the Usual Management With or Without Physical Training
Acronym: FRAM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not be set up due to recruitment and feasibility problems
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GREMEAUX PHRC I 2015
Record Dates: First submitted 2017-08-04; First posted 2017-08-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual management (Other)
  Interventions: Other: no physical activity
- physical training (Experimental)
  Interventions: Other: physical activity

INTERVENTIONS:
Other: no physical activity — no physical activity
  Arms: usual management
Other: physical activity — Rehabilitation program will start 4 weeks after discharge from acute care (S4), for a duration of 8 weeks (3 sessions / week). Physical training will include aerobic exercises 30-60 minutes at 50-80% of HRmax, associated with muscle building exercises in circuit training (20 min), and balance and flexibility exercises.
  Arms: physical training

SUMMARY:
After a minor stroke, patients frequently report complaints such as fatigue and difficulty with certain everyday motor tasks, leading to a marked deterioration in their quality of life. The aim of this study is to show that the implementation of a personalised physical activity programme, starting 1 month after the hospitalisation for minor stroke, significantly decreases the frequency of fatigue in these patients, in comparison with usual management "in real life"..

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* National health insurance cover
* 1st minor ischaemic stroke (initial NIH score ≤ 4)
* Satisfactory neurological recovery at discharge from hospital (modified Rankin score ≤2)
* Patient living close to the participating centre (<50 km)
* With early post-stroke fatigue (FFS score ≥ 4 at the definitive inclusion visit (W3))

Exclusion Criteria:

* haemorrhagic stroke
* History of ischaemic or haemorrhagic stroke with clinical manifestations
* History of TIA
* MMS ≤ 24
* Pre-existing dementia (defined according to DSM IV criteria)
* Neurosensory or orthopaedic disorders requiring permanent technical support before the stroke and making reconditioning impossible
* Aggravation of the neurological status after the initial hospitalisation (NIH score ≥ 6)
* Recurrence of the cerebrovascular event or onset of an acute cardio-vascular event between the screening and definitive inclusion
* Pre-stroke Rankin score ≥ 3
* Pregnant patient
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Fatigue relief (assessed by the Fatigue Severity Scale) | 4 months after the stroke

REFERENCES:
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300